CLINICAL TRIAL: NCT02247583
Title: Investigating Patient Satisfaction With Oral Anti-Cancer Treatment. Prospective Non-interventional Non-controlled Multicenter Observational Study to Evaluate Aspects of Pharmaceutical Care in Patients With Advanced Renal Cell Carcinoma Treated With an Oral Anti-cancer Drug.
Brief Title: Investigating Patient Satisfaction With Oral Anti-Cancer Treatment
Acronym: IPSOC
Status: Completed | Type: Observational
Sponsor: KU Leuven (Other)
Collaborators: Flemish League Against Cancer (Other); Pfizer (Industry); Novartis (Industry); GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Sandra De Coster, Pharmacist, KU Leuven
Other Study IDs: VF/2010/03; s52586 (Registry Identifier: Clinical Trial Center UZ Leuven)
Record Dates: First submitted 2014-07-03; First posted 2014-09-25 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Clear Cell Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- mRCC patients: Patients with metastatic renal cell carcinoma

SUMMARY:
Prospective non-interventional non-controlled multicenter observational study to evaluate aspects of pharmaceutical care in patients with advanced renal cell carcinoma treated with an oral anti-cancer drug.

The main objective of this study is to evaluate the patient perspective in the treatment of advanced renal cell carcinoma with an oral anti-cancer drug.

The following aspects will be investigated:

* Intrinsic desire for information about treatment.
* Patient satisfaction with treatment information.
* Patient satisfaction with treatment.
* Medication adherence.
* Health-related quality of life.
* The role of different health care professionals in the treatment of RCC with oral drugs

This study should reveal information necessary for the development of pharmacotherapeutic care concepts that meet the needs of cancer patients treated with an oral anti-cancer drug over a long period.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are 18 years or older, and who can be contacted by phone and/or e-mail are eligible for the study

Exclusion Criteria:

* Patients who are not able to understand Dutch or French will be excluded from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: mRCC patients starting with an oral anti-cancer treatment
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2011-02; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Medication adherence | one year
  At the first visit patients will receive their anti-cancer medication by the hospital in a pill box which electronically records openings cf. Medication Event Monitoring System (MEMS®, Aardex). The recorded information in this chip will be read in the hospital pharmacy each time the patient gets new capsules. This information is strictly confidential and can only be consulted by the research team at the KULeuven.

SECONDARY OUTCOMES:
Extent of Information Desire (EID) | one year
  Extent of information desire will be assessed, using a standardised questionnaire, at the start of the treatment, after approximately 1, 3 and 6 months of treatment and after about 12 months, at discontinuation of therapy or at end of study (whatever is earlier).
Patient Satisfaction with Cancer Treatment Education (Ps-CaTE) | one year
  Satisfaction with cancer treatment information will be assessed, using a standardised questionnaire, after approximately 1, 3 and 6 months of treatment and after about 12 months, at discontinuation of therapy or at end of study (whatever is earlier).
Morisky Medication Adherence Scale (MMAS) | one year
  Medication adherence will be assessed, using a standardised questionnaire, after approximately 1, 3 and 6 months of treatment and after about 12 months, at discontinuation of therapy or at end of study (whatever is earlier).
Cancer Therapy Satisfaction Questionnaire (CTSQ) | one year
  Satisfaction with cancer treatment will be assessed, using a standardised questionnaire, after approximately 1, 3 and 6 months of treatment and after about 12 months, at discontinuation of therapy or at end of study (whatever is earlier).
Functional Assessment of Cancer Therapy - General (FACT-G) | one year
  Health-related quality of life will be assessed, using a standardised questionnaire, at the start of the treatment, after approximately 1, 3 and 6 months of treatment and after about 12 months, at discontinuation of therapy or at end of study (whatever is earlier).
Functional Kidney Symptom Index (FKSI) | one year
  Health-related quality of life will be assessed, using a standardised questionnaire, after approximately 1, 3 and 6 months of treatment and after about 12 months, at discontinuation of therapy or at end of study (whatever is earlier).
Satisfaction With Pharmacist (SwiP) | one year
  Satisfaction with the pharmacist will be assessed, using a standardised questionnaire, after approximately 1, 3 and 6 months of treatment and after about 12 months, at discontinuation of therapy or at end of study (whatever is earlier).

CONTACTS AND LOCATIONS:
Overall Officials: Veerle Foulon, Professor, Study Director — Katholieke Universiteit Leuven - Klinische Farmacologie en Farmacotherapie
Locations (1):
- Katholieke Universiteit Leuven - Klinische Farmacologie en Farmacotherapie, Leuven, Belgium